CLINICAL TRIAL: NCT06570902
Title: Prospective WCD Post CABG Registry
Brief Title: Prospective WCD Post CABG Registry (CABG Registry)
Status: Recruiting | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0270
Record Dates: First submitted 2024-07-28; First posted 2024-08-26 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Cardiomyopathy Ischemic; Cardiomyopathies; Cardiovascular Diseases; Heart Disease, Ischemic
MeSH Terms: conditions — Cardiomyopathies; Cardiovascular Diseases; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: WCD — An FDA-approved, CE marked WCD will be prescribed for up to 3 months of use after hospital discharge, with the option for longer use under physician discretion

SUMMARY:
The primary objective is to observe the rate of recovery of ventricular function (EF>35%) after first-time coronary artery bypass graft surgery in patients who were prescribed the wearable cardioverter defibrillator (WCD) post-surgery prior to being discharged after hospitalization as part of standard clinical care.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the rate of recovery of ventricular function (EF>35%) in patients with ischemic heart failure with reduced ejection fraction (EF ≤35%) after undergoing first time, coronary artery bypass grafting (CABG) procedure while being treated with guideline-directed medical therapy (GDMT). It is anticipated that more patients will have EF recovery as compared to a retrospective register where 54% of isolated CABG patients had EF recovery by end of WCD use (Kuehn et al., 2022), mostly driven by the modern improved usage of GDMT drugs.

This study is designed as a multi-center prospective observational study of patients who underwent first time coronary artery bypass grafting procedure with HFrEF at hospital discharge to test the hypothesis that EF recovery will be improved by end of WCD wear due to increased usage of GDMT. The study will target 20% female enrollment and recruitment will be adjusted if the percentage of female subjects enrolled are far from 20%.

ELIGIBILITY:
Inclusion Criteria

* Patient underwent first-time CABG surgery <10 days before enrollment.
* Patient is prescribed WCD for a primary reason of HF with reduced EF < 35% measured after surgery but before hospital discharge.
* Patient is ≥18 years old

Exclusion Criteria:

* Patients having combination CABG surgery with heart valve repair.
* Patients with prior CABG.
* Patients who have an active unipolar pacemaker.
* Patients with a physical or mental condition that could impair their ability to properly interact with the WCD.

Patients currently participating in an interventional clinical study. Patients with any skin condition that would prevent wearing the device. Patients with an advanced directive prohibiting resuscitation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were prescribed the wearable cardioverter defibrillator (WCD) post-surgery prior to being discharged after hospitalization as part of standard clinical care
Sampling Method: Probability Sample
Enrollment: 910 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
EF recovery | Enrollment till WCD End of Use
  EF recovery at end of WCD use, usually after 90days of wear. End of WCD use will be determined by the prescribing physician. For this study, EF>35% will be considered as EF recovery.

SECONDARY OUTCOMES:
Quality of Life (KCCQ | Enrollment till WCD End of Use, usually up to three month
  Quality of Life (QoL) information will be collected using the following questionnaires:
  - Kansas City Cardiomyopathy Questionnaire short form (KCCQ-12)
Quality of Life EQ | Enrollment till WCD End of Use, usually up to three month
  Quality of Life (QoL) information will be collected using the following questionnaires:
  - EQ-5D-5L
Medication Adherence | Enrollment till WCD End of Use, usually up to three month
  Medications and self-reported adherence to taking those medications as prescribed will be recorded from chart review and patient interview, if necessary, every month (30 days). Medications will also be recorded at the start and end of WCD use
Healthcare utilization | Enrollment till WCD End of Use, usually up to three month
  Information (days, reasons) on any hospitalizations, emergency room visits, observation stays, urgent care visits, other physician office visits, and stays at skilled nursing facilities.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Kerckhoff Klinik, Bad Nauheim, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Sana-Herzzentrum Cottbus GmbH, Cottbus
  - Universitätsklinikum Halle (Saale), Halle

IPD SHARING:
Plan to Share IPD: Undecided